CLINICAL TRIAL: NCT06513897
Title: The Effects of Acupressure and Paternal Holding on Pain and Physiological Parameters in Infants During Heel Lancing: a Randomized Controlled Trial
Brief Title: The Effects of Acupressure and Paternal Holding on Pain and Physiological Parameters During Heel Lancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Ilcim Ercan Koyuncu, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Heel Lancing
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-07

CONDITIONS: Infant Development; Nurse's Role; Pain, Acute
Keywords: acupressure; heel lancing; infant; father's lap
MeSH Terms: conditions — Acute Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupressure (Experimental)
  Interventions: Other: Acupressure
- Paternal Holding (Experimental)
  Interventions: Other: Father's Lap
- Control (No Intervention)

INTERVENTIONS:
Other: Acupressure — Acupressure will be applied to the foreheads of the babies in this group starting two minutes before the heel prick. Acupressure application will be finished when heel prick blood collection is finished.
  Arms: Acupressure
Other: Father's Lap — Infants in this group will be placed on the father's lap two minutes before heel prick blood collection. They will remain on the father's lap during the heel prick procedure.
  Arms: Paternal Holding

SUMMARY:
Neonatal heel blood collection is a common medical procedure to obtain blood samples from newborns for diagnostic purposes. Although necessary for clinical evaluation, this procedure causes discomfort and distress in infants. The pain experienced during heel prick is a major concern and warrants exploration of effective and compassionate interventions to alleviate associated discomfort and reduce crying time. Non-pharmacological approaches, such as acupressure and cuddling, are thought to have important contributions to improving the overall experience of newborns undergoing this procedure. . The aim of this study was to evaluate the efficacy of acupressure and paternal hugging interventions in relieving pain and reducing crying time during neonatal heel haemorrhage. The choice of these interventions was based on their potential to offer non-invasive and holistic approaches to pain management by addressing not only the physical but also the emotional dimensions of the neonatal experience.

DETAILED DESCRIPTION:
Neonatal heel prick blood collection is a common medical procedure performed to obtain blood samples from newborns for diagnostic purposes. Neonatal heel prick plays an important role in the diagnosis of genetic and metabolic diseases such as hypothyroidism and phenylketonuria. Although necessary for clinical evaluation, this procedure causes discomfort and distress in infants. Pain during heel prick is a major concern and warrants exploration of effective and compassionate interventions to alleviate the associated discomfort and reduce crying time. In this sense, there are studies on both heel prick instruments and interventions applied to the infant during heel prick. Non-pharmacological approaches such as acupressure and hugging are thought to have important contributions to improving the overall experience of newborns undergoing this procedure. It is known that one of the most important determinants of attachment in the postnatal period is touch, hugging and skin-to-skin contact. The neonatal period is a critical developmental stage characterised by rapid physiological and neurological changes. It is thought that the sensitivity of newborns to pain and early painful experiences may have potential long-term effects. There are studies suggesting that painful procedures may be effective in mother-baby or father-baby attachment. While there are studies in the literature on mother's hug, no study on father's hug was found. Due to the role of the presence of fathers in paediatric pain management, the potential to provide emotional support, the father's hug as a form of comforting touch, contributing to the release of oxytocin, a hormone associated with attachment and stress reduction, and the emotional bond established through hugging may act as a buffer against distress associated with painful procedures and promote a sense of security and assurance in the infant, it was considered appropriate to use it in this study. Acupressure, derived from traditional Chinese medicine, involves applying manual pressure to specific points on the body to promote healing and relieve pain. Similarly, emotional support provided by a carer, such as a father, through cuddling is thought to have the potential to reduce stress and improve the infant's emotional well-being. In this study, investigators aimed to evaluate the effectiveness of acupressure and paternal hug interventions in relieving pain and reducing crying time during neonatal heel haemorrhage. The choice of these interventions was based on their potential to offer non-invasive and holistic approaches to pain management by addressing not only the physical but also the emotional dimensions of the neonatal experience.

ELIGIBILITY:
Inclusion Criteria:

* Being a term newborn
* A healthy newborn with its mother by its side
* Not taking any analgesic/sedative medication within 24 hours
* The baby has not undergone invasive procedures other than routine interventions

Exclusion Criteria:

* Preterm-postterm newborn
* Having a systemic disease
* Taking analgesic/sedative medication in the last 24 hours
* Invasive procedures other than routine interventions

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Pain Score | pre-intervention, immediately after the intervention
  Pain will be assessed using the Neonatal Pain, Agitation, Sedation Scale. The minimum score of the scale is 0 and the maximum score is 10. Four points and below is considered as mild pain, five points and above is considered as moderate and severe pain.
Pulse value | pre-intervention, immediately after the intervention
  Pulse value will be assessed using the infant pulse oximeter.
Crying time | During the intervention
  Crying time will be recorded throughout the procedure.
Saturation value | pre-intervention, immediately after the intervention
  Saturation value will be assessed using the infant pulse oximeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoarau K, Payet ML, Zamidio L, Bonsante F, Iacobelli S. "Holding-Cuddling" and Sucrose for Pain Relief During Venepuncture in Newborn Infants: A Randomized, Controlled Trial (CASA). Front Pediatr. 2021 Jan 14;8:607900. doi: 10.3389/fped.2020.607900. eCollection 2020. PMID 33520895
- [Background] Devi R, Priyadarshi M, Singh P, Chaurasia S, Basu S. Neonatal Pain Response to Various Heel Prick Devices: A Randomized Controlled Trial. Indian Pediatr. 2023 Nov 15;60(11):893-898. Epub 2023 Jun 21. PMID 37551876
- [Background] Adeli M, Aradmehr M. A comparative study of maternal-neonate abdominal and kangaroo (skin-to-skin) skin contact immediately after birth on maternal attachment behaviors up to 2 months. J Educ Health Promot. 2018 Mar 1;7:42. doi: 10.4103/jehp.jehp_46_16. eCollection 2018. PMID 29619393
- [Background] Abraham E, Hendler T, Shapira-Lichter I, Kanat-Maymon Y, Zagoory-Sharon O, Feldman R. Father's brain is sensitive to childcare experiences. Proc Natl Acad Sci U S A. 2014 Jul 8;111(27):9792-7. doi: 10.1073/pnas.1402569111. Epub 2014 May 27. PMID 24912146